CLINICAL TRIAL: NCT05413694
Title: Epidemiological Monitoring of COVID-19 Patients Hospitalized on Reunion Island
Acronym: COVIDEPI-SUIV'
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/CHU/04
Record Dates: First submitted 2022-06-09; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- telephone interview 24 months after hospitalization for Covid-19 (Experimental): telephone interview 24 months after hospitalization for Covid-19
  Interventions: Other: telephone interview 24 months after hospitalization for Covid-19

INTERVENTIONS:
Other: telephone interview 24 months after hospitalization for Covid-19 — telephone interview 24 months after hospitalization for Covid-19

SUMMARY:
The island of Reunion, a French overseas department of 860,000 inhabitants, located in the Indian Ocean (OI) zone, recorded its first case of COVID-19 on March 11, 2020. The epidemic, which was described as not very severe during the year 2020 in Reunion was much more intense and more deadly in 2021, with the arrival of the new variants (South African and Indian) and exploded at the beginning of the year 2022 (variant Omicron).

Reunion has a specific island context both climato-geographically and demographically. Indeed, this French island located in the southern hemisphere in the middle of the Indian Ocean (OI) has a tropical climate and a multi-ethnic population, younger than in mainland France (16% are over 60 years old). It is also marked by a higher prevalence in the general population of certain risk factors, such as obesity (11%) and type 2 diabetes (>10%), recognized as factors favoring severe clinical forms of COVID-19. as well as "persistent COVID-19".

This study will allow the constitution of a large-scale French cohort located in a closed overseas territory to provide answers to local specificities and to the management of the epidemic in the territory.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* having been hospitalized at the University Hospital Center (CHU) of Reunion (minimum of one night in the hospital)
* with a positive diagnosis of COVID-19 (positive RT(reverse transcription)-PCR(Polymerase Chain Reaction) SARS-CoV-2 on a nasopharyngeal swab or positive serology or confirmed diagnosis in the medical file)
* registered in the COVIDEPI database
* whose telephone numbers are available in the computerized patient file
* residing on the island of Reunion
* knowing how to understand and speak French

Exclusion Criteria:

* deceased
* opposing the use of their data
* deprived of liberty by judicial or administrative decision, minors, and persons subject to a legal protection measure: guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of patients with "persistent COVID-19" | 24 month
  presence (at the time of the interview or in the month preceding the interview) of at least one symptom among the most frequent prolonged symptoms of COVID-19 and which was not present before the interview SARS (severe acute respiratory syndrome )-CoV-2 infection

SECONDARY OUTCOMES:
Determine the factors associated with the persistence of symptoms | 24 month
Measure physical and mental quality of life | 24 month
  Medical Outcome Study Short Form 12

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No